CLINICAL TRIAL: NCT05122013
Title: A Comprehensive Remote Intervention Program for Weight Regain After Sleeve Gastrectomy: An Open Label Randomized Controlled Trial
Brief Title: Remote Intervention for Weight Regain After Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Dr Shiri Sherf-Dagan (RD, PhD) Dietitian and Epidemiologist, Principal Investigator, Assuta Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0046-21-ASMC
Record Dates: First submitted 2021-10-19; First posted 2021-11-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: Bariatric Surgery; Weight gain; Telemedicine
MeSH Terms: conditions — Obesity; Weight Gain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be recruited to the study and randomized to intervention or control group. Medical and demographic data collection as well as measurements and validated questionnaires will be conducted at baseline (T0) and after the intervention (3 months after T0). In addition, at 3- and 6-months post intervention patients will be contacted via phone calls and asked about their weight, physical activity, sleeping and nutritional habits, and adherence to bariatric surgery recommendations. At T0, the intervention group will be scheduled for remote meetings and the the control group will receive a single meeting with the study's registered dietitian at the end of data collection of T0, along with a recommendation to continue follow-up and lifestyle changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Other): The comprehensive 3-month remote intervention program by the multidisciplinary study team includes 6-weeks of online meetings with the study registered dietitian, sleep and physical activity consultants, followed by another 6-weeks of online meetings with the study's registered dietitian, overall 12 weeks containing a total of 12 remote consultations (6 dietitian, 3 physical activity consultant, 3 sleep consultant). In addition, the intervention group will receive weekly text messages to their mobile phone, meant to enhance happiness and subjective wellbeing.
  Interventions: Behavioral: A comprehensive remote multidisciplinary intervention for weight regain after sleeve gastrectomy
- control group (Other): The control group will receive standard nutrition care: A one-time meeting with the study's registered dietitian at the clinic, focusing on nutrition and behavioral recommendations, followed by the standard recommendation to continue follow up, engage in physical activity and general lifestyle recommendations.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: A comprehensive remote multidisciplinary intervention for weight regain after sleeve gastrectomy — A remote 3-months multidisciplinary intervention for weight regain after sleeve gastrectomy including bi-monthly remote consultations with a registered dietitian, physical activity consultant and sleep consultant, combined with weekly text messages meant to enhance happiness and subjective wellbeing.
  Arms: intervention group
Behavioral: Control group — Standard nutritional care: One frontal meeting with the study's registered dietitian at the clinic, including nutritional and behavioral assessment and recommendations, followed by guidance to to continue follow up in order to support healthy lifestyle.
  Arms: control group

SUMMARY:
The study is designed to assess the effect of a 3-month remote comprehensive intervention program by a multidisciplinary team combined with mobile supportive text messages aimed to raise the level of happiness and subjective wellbeing, on weight outcomes and physical and behavioral parameters among bariatric surgery patients after sleeve gastrectomy who had a weight regain of ≥10% from nadir, compared to a control group which will receive standard care of a single meeting with the study's registered dietitian at the clinic and then be advised to continue follow up.

DETAILED DESCRIPTION:
One hundred patients will be recruited to the study and randomized to intervention or control group. The comprehensive 3-month remote intervention program by the multidisciplinary study team includes 6-weeks of online meetings with the study registered dietitian, sleep and physical activity consultants, followed by another 6-weeks of online meetings with the study RD, overall 12 weeks containing a total of 12 remote consultations (6 dietitian, 3 physical activity consultant, 3 sleep consultant). In addition, the intervention group will receive weekly text messages to their mobile phone, meant to enhance happiness and subjective wellbeing.

The control group will receive standard care of a single meeting with the study's registered dietitian at the clinic including nutrition and behavioral recommendations and then advised to continue follow up, engage in physical activity and general lifestyle recommendations.

Both groups will undergo comprehensive tests at baseline and at the end of intervention after 3 months. Patients from both groups who will arrive to the follow-up appointment after 3 months will receive a participation reward which will include a gift card on the sum of 154 NIS for purchasing a multivitamin package for bariatric patients.

Finally, 3 and 6 months after intervention completion, self-reported data will be collected via phone calls including weight, physical activity (type, times per week and duration per time), professional follow up and adherence to BS recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age at the time of BS ≥18 years
* Patients who underwent primary SG at least 2 years ago and regained at least 10% weight from nadir.
* Read and speak Hebrew.

Exclusion Criteria:

* Patients who underwent more than one BS in their past.
* Use of weight loss drug therapy currently or 1-month prior to trial entry.
* Currently attending a weight loss program and lost more than 5% of weight at the last month.
* Current pregnancy and women who gave birth in the last 6 months.
* Medical contraindications such as active cancer, organ transplant or unbalanced psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
The effect of a comprehensive remote multidisciplinary intervention program focused on weight regain after sleeve gastrectomy on weight change, compared to a control group. | Changes from baseline at 3 months
  Weight change in kilograms will be measured before and at the end of the 3-month intervention, for both intervention and control group.

SECONDARY OUTCOMES:
The effect of the intervention on behavioral recommendations. | Changes from baseline at 3, 6, and 9 months
  Compliance to bariatric surgery recommendations will be assessed before and at the end of the 3-month intervention, and also 3 and 6 months after the intervention has ended, for both intervention and control group, each time regarding the last month. Patients will be asked if they currently keep the main recommended bariatric surgery behaviors in the last month (0-never done, 1-partially done, 2-always done).
The effect of the intervention on grazing. | Changes from baseline at 3 months
  Grazing will be assessed before and at the end of the 3-month intervention, for both intervention and control group, by using two questions from the grazing questionnaire by lane et al: "Do you graze between meals?" and "would you describe the way you generally eat as unplanned and repetitious (i.e. eating between planned meals and snacks)?", each time regarding the last month. Answering Yes for 1 or 2 of the questions will be considered as grazing behaviour.
The effect of the intervention on food tolerance. | Changes from baseline at 3 months
  Food tolerance will be assessed before and at the end of the 3-month intervention, for both intervention and control group, by asking the patients "regarding the last month, Are there any types of foods or beverages that you cannot eat because of intolerance (suffering from pain or discomfort after eating a small amount)?". This question was based on the validated questionnaire by Suter et al. an answer of yes will indicate food intolerance, the more foods and drinks detailed the worse the intolerance is.
The effect of the intervention on subjective binge eating. | Changes from baseline at 3 months
  Subjective binge eating habits will be assessed before and at the end of the 3-month intervention, for both intervention and control group. Patients will be asked it they have had episodes of eating subjectively large amounts of food while experiencing a sense of loss of control at least once a week in the last 3 months, according to the DSM-5 definition.
The effect of the intervention on dietary intake by food diaries. | Changes from baseline at 3 months
  Dietary intake will be assessed before and at the end of the 3-month intervention, for both intervention and control group. Patients will be asked to fill food diaries for 3 days consisting of 2 week days and 1 weekend day. Daily average intake in calories will be calculated based based on the "Nutratio" software.
The effect of the intervention on dietary intake by 24-hour recall. | Changes from baseline at 3 months
  Dietary intake will also be assessed before the intervention, for both intervention and control group, by a 24-hour dietary recall. To reduce information bias, patients will be shown examples of standard cups, spoons, teaspoons and foods using the Israeli food atlas and visual measuring tools. Daily average intake in calories will be calculated based on the "Nutratio" software.
The effect of the intervention on dietary intake by food frequency questionnaire (FFQ). | Changes from baseline at 3 months
  Dietary intake will also be assessed before the intervention, for both intervention and control group, by a FFQ. To reduce information bias, patients will be shown examples of standard cups, spoons, teaspoons and foods using the Israeli food atlas and visual measuring tools. Daily average intake in calories will be calculated based on the "Nutratio" software.
The effect of the intervention on food environment's impact on eating behaviors. | Changes from baseline at 3 months
  Food environment's impact on eating behaviors will be assessed before and at the end of the 3-month intervention, for both intervention and control group, by a validated questionnaire "Power of food scale". Each of the 15 questions gets a score between 0 (Do not agree at all) to 5 (strongly agree). The scores are summed up between 0-75, a higher score indicating higher sensitivity to food environment.
The effect of the intervention on physical activity habits. | Changes from baseline at 3, 6, and 9 months
  Patients will be asked at baseline and at the end of the intervention program about their physical activity regimen including type, duration of each session and times per week. In addition, self-reported physical activity levels will be collected via phone calls at 3 and 6 months after the end of the intervention program. Data of minutes of physical activity per week will be compared between groups.
The effect of the intervention on functionality regarding upper extremity strength. | Changes from baseline at 3, 6, and 9 months
  Strength of the upper extremities will be measured before and at the end of the 3-month intervention program, for both intervention and control group, by a digital hand dynamometer (Jamar plus digital). Measurements will be taken three times for the dominant hand with a break of 15 seconds between each measurement, and an average will be calculated. Results in kilograms will be compared to manufacturer's normal values by age and gender.
The effect of the intervention on functionality regarding lower extremity strength . | Changes from baseline at 3, 6, and 9 months
  To assess lower extremity strength, the 5 times sit and stand test will be used before and at the end of the 3-month intervention program, for both intervention and control group. Time in seconds to complete the test will be measured, faster time indicating better lower extremity strength.
The effect of the intervention on sleeping habits. | Changes from baseline at 3 months
  Sleeping quality will be assessed before and at the end of the 3-month intervention for both intervention and control group, each time regarding the last month, by a validated questionnaire - The Pittsburgh Sleep Quality Index (PSQI).The PSQI includes 19 questions grouped into components, each on a 0-3 point scale. Scores of >5 indicate subjective insomnia. Moreover, 3 and 6 months after the end of the intervention complement, patients from both intervention and control group will be asked by phone call about their average sleeping hours on weekdays and weekends.
The effect of the intervention on sleeping hours. | Changes from baseline at 3 months
  Three and 6 months after the end of the intervention complement, patients from both intervention and control group will be asked by phone call about their average sleeping hours on weekdays and weekends.
The effect of the intervention on happiness and subjective wellbeing | Changes from baseline at 3, 6, and 9 months
  Happiness and subjective wellbeing will be assessed before and at the end of the 3-month intervention for both intervention and control group using a structured questionnaire by Sherman and Shavit. The questions include patients subjective well-being by asking them to assess their present life on a Likert-type scale from 0 representing "worst possible life" to 10 representing "best possible life".
The effect of the intervention on weight 3 and 6 months after the end of the intervention. | Changes from baseline at 3, 6, and 9 months
  Self-reported weight in kilograms at 3 and 6 months after the intervention complement will be asked by phone call for both intervention and control group.
The effect of the intervention on attendance to follow up meetings 3 and 6 months after the end of the intervention. | Changes from baseline at 3, 6, and 9 months
  Self-reported number of follow up meetings at 3 and 6 months after the intervention complement will be asked for both intervention and control group. Patients will be asked how many meetings they had with a registered dietitian, a psychologist/social worker, a surgeon and a personal trainer.
The effect of the intervention on supplementation usage 3 and 6 months after the end of the intervention. | Changes from baseline at 3, 6, and 9 months
  Self-reported supplementation usage at 3 and 6 months after the intervention complement will be asked for both intervention and control group regarding the last month.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No